CLINICAL TRIAL: NCT06446817
Title: Multicentric Clinical Investigation to Determine Safety and Efficacy of a Hydrophobic Acrylic Multifocal Intraocular Lens
Brief Title: Bicentric Clinical Investigation to Assess Safety and Performance of LuxHighAdd IOL
Acronym: HIGHADD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cutting Edge SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE2301; 2023-A01904-41 (Registry Identifier: French BRC Identification number)
Record Dates: First submitted 2024-05-23; First posted 2024-06-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LuxHighAdd (Experimental): The experimental group will recieve the LuxHighAdd intraocular lens bilaterally.
  Interventions: Device: LuxHighAdd IOL
- LuxGood group (Active Comparator): The control group will recieve the LuxGood intraocular lens bilaterally.
  Interventions: Device: LuxGood IOL

INTERVENTIONS:
Device: LuxHighAdd IOL — Bilateral implantation in the capsular bag to replace the cataractous human crystalline lens.
  Arms: LuxHighAdd
Device: LuxGood IOL — Bilateral implantation in the capsular bag to replace the cataractous human crystalline lens.
  Arms: LuxGood group

SUMMARY:
The study purpose is to demonstrate safety and performance of bilateral implantation of LuxHighAdd intraocular lens compared with the LuxGood Monofocal lens.

DETAILED DESCRIPTION:
The study purpose is to demonstrate safety and performance after bilateral implantation of LuxHighAdd intraocular lenses.

The device under investigation is a hydrophobic acrylic multifocal intraocular lens (IOL) manufactured by the sponsor of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 50 or over on the day of inclusion, presenting a bilateral cataract, qualified for bilateral implantation
* No ocular comorbidity possibly affecting the study results
* Fit within the available IOL diopter range
* Have had no previous refractive surgery
* Regular corneal astigmatism ≤1.0 dioptres
* Clear intraocular media other than cataract
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Ability to attend all study follow-ups
* Signed informed consent.

Exclusion Criteria:

* Ocular surface disease potentially affecting study results
* Pre-existing ocular pathology or history of pathology potentially affecting the study results
* Acute or chronic disease or illness that would increase risk or confound study results
* Subjects who may be reasonably expected to require a secondary surgical intervention at any time during the investigation (other than YAG capsulotomy)
* Axial lengths and keratometry such as the IOL spherical power is not in the range of 16 to 26 D
* Instability of keratometry or biometry measurements
* Traumatic cataract
* Amblyopia
* History of ocular trauma or any prior ocular surgery including refractive procedures
* Capsular or zonular abnormalities that may affect postoperative centration or tilt of the lens
* Pupil abnormalities
* Systemic or ocular medication that could modify pupil dynamics
* Expected complicated surgery or complicated surgery
* Concurrent participation in another drug or device investigation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Distance Corrected Near Visual Acuity (DCNVA) | 4/6 months after surgery
  To demonstrate the difference in monocular DCNVA between the High Add lens and the LuxGood monofocal lens by means of statistical significance.
Best corrected distance visual acuity (BCDVA) | 4/6 months after surgery
  To demonstrate the non-inferiority of the Lux High Add lens compared with the monofocal control LuxGood lens in terms of BCDVA by means of statistical significance.

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | 4/6 months after surgery
  Uncorrected photopic visual acuity at far in monocular and binocular with LuxHighAdd lens compared to LuxGood lens.
Uncorrected Intermediate Visual Acuity (UIVA) | 4/6 months after surgery
  Uncorrected photopic visual acuity at intermediate distance in monocular and binocular with LuxHighAdd lens compared to LuxGood lens.
Uncorrected Near Visual Acuity (UNVA) | 4/6 months after surgery
  Uncorrected photopic visual acuity at near distance in monocular and binocular with LuxHighAdd lens compared to LuxGood lens.
Distance Corrected Intermediate Visual Acuity (DCIVA) | 4/6 months after surgery
  Photopic visual acuity at intermediate distance in monocular and binocular with best distance correction with LuxHighAdd lens compared to LuxGood lens.
Manifest Refraction | 4/6 months after surgery
  Manifest subjective refraction
Defocus curve | 4/6 months after surgery
  Binocular defocus curve with the distance correction
Adverse events rates | 4/6 months after surgery
  Adverse events rates
Contrast Sensitivity | 4/6 months after surgery
  Contrast Sensitivity in binocular conditions with distance correction
Halo and glare scores | 4/6 months after surgery
  Halos and glare assessed with a simulator
Patient-reported outcomes: Quality of vision Questionnaire | 4/6 months after surgery
  Assessment of quality of vision (CatQuest-9SF)
Patient-reported outcomes: Spectacle independance Questionnaire | 4/6 months after surgery
  Assessment of spectacle independence (PRSIQ questionnaire )
Patient-reported outcomes: open-ended question | 4/6 months after surgery
  Frequency and proportion of eyes with ocular and visual symptoms (non-directed complaints) using an open-ended question

CONTACTS AND LOCATIONS:
Overall Officials: Alain Saad, MD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (2):
- France (2):
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - WestOphta, Rennes